CLINICAL TRIAL: NCT05958758
Title: An Open Label Pragmatic Feasibility Study on a Resilience Focused Community of Practice Program With Psilocybin-assisted Therapy (PaT) for End-of-Life Patients.
Brief Title: A Community of Practice Program With Psilocybin-assisted Therapy for End-of-Life Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Roots to Thrive Society for Psychedelic Therapy (Other)
Collaborators: Vancouver Island Health Authority (Other); Vancouver Island University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H22-02523
Record Dates: First submitted 2023-02-23; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: End of Life
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Group administered Psilocybin-assisted therapy
  Interventions: Drug: Psilocybin-assisted therapy within a community of practice model (group administered)

INTERVENTIONS:
Drug: Psilocybin-assisted therapy within a community of practice model (group administered) — The community of practice is 10 weeks long, meeting virtually for 2 hours each week, in a structured process, run through the Roots to Thrive treatment program. The psilocybin-assited therapy sessions occur midway through the 10-week program.

SUMMARY:
The purpose of the study is to understand the feasibility of a resilience focused community of practice program that includes psilocybin-assisted therapy for End-of-Life Distress. The community of practice refers to a research informed group therapy process that runs over a 10-week period of time and includes one group administered psilocybin-assisted therapy session.

Target population: The treatment team will treat a total of 64 patients who have:

* a terminal diagnosis (experiencing end of life distress),
* AND who are eligible for the RTT + Psilocybin-assisted Therapy Treatment program through the RTT Society.

DETAILED DESCRIPTION:
Treatment will take place at the Snuneymuxw Traditional Medicines Clinic, 1984 Woobank Rd, Nanaimo, B.C.Research data will be coordinated and held through RedCap, hosted by Island Health.

Data collection centres on 1) understanding the feasibility; 2) collecting safety data; 3) exploring the mental health impacts of a community of practice as the vessel for psilocybin-assisted therapy for those with end-of-life distress.

There is a mixed method approach for data collection, including:

* Collect attendance
* Biomedical measures taken during psilocybin sessions (blood pressure, pulse, medications to manage side effects).
* Quantitative Health and Wellness Questionnaires of participants before, within, immediately after, and six months after completion.
* Qualitative Surveys and Exit Interviews.

ELIGIBILITY:
Inclusion Criteria

* Patient must have a terminal diagnosis whereby there is a limited life expectancy (predicted life expectancy less than 2 years).
* Ages 19-80 years of age
* Male, menopausal female, if childbearing age not pregnant, using birth control and negative pregnancy test prior to psilocybin administration.
* Ambulatory (Palliative performance status 50% or greater)
* eGFR >20 ml/min ❏AST < 3xULN and bilirubin <50 umol/L
* Patient has emotional distress that has not successfully responded to other treatments: other treatments failed, patient could not tolerate other treatments, patient is unable to access other treatments, or patient refused other treatments for reasons acceptable to our treatment team.
* Patient demonstrates comprehension sufficient for understanding the consent form.

Exclusion Criteria:

* Treatment in a clinical trial where psilocybin therapy would disqualify them from their primary treatment trial.
* If female is:a) pregnant (positive pregnancy test),b) nursing,
* Currently taking on a regular (e.g., daily) basis: >investigational agents, >medications that are MAO inhibitors >UDG modulators, and inhibitors of UGT1A9 and 1A10, aldehyde or alcohol dehydrogenase inhibitors, SSRI's, SNRI's.

  * Patients are given the option to wean themselves off their medications prior to the psilocybin to be included in the trial. Patients taking MAO-A inhibitors (especially the irreversible inhibitors) will require a minimum 2-week washout period. The possible concern over serotonin syndrome with these agents is not well documented in the literature, however the long interval before MAO is replenished may warrant a cautious approach based on the patient's risk factors and warrants oversight from the MRP (Most Responsible Physician)
  * Patientstaking MAO-B inhibitors should be assessed on a case by case basis as there is a potential for a heightened response and warrants oversight from the MRP.
* Patients with known sensitivities to psilocybin and or its metabolites or have had significant adverse events after prior psilocybin or other psychedelic use.
* Active uncontrolled epilepsy.
* Uncontrolled cardiovascular conditions: uncontrolled hypertension, uncontrolled angina, a clinically significant ECG abnormality (e.g. QT prolongation).
* Uncontrolled vascular disease (such as TIA in the last 3-6 months, stroke with loss in mental status, peripheral or pulmonary vascular disease with active claudication).
* Unstable Insulin-dependent diabetes;

Conditions requiring special medical consideration:

* Cancer has central nervous system involvement.
* Paraneoplastic syndrome or a tumor with ectopic hormone production which may place the patient at risk for hypercalcemia, Cushing's syndrome, or SIADH secretion.

Psychiatric Exclusion Criteria:

* Severity of depression or anxiety symptoms warranting immediate emergent treatment with antidepressant or daily anxiolytic medication as these patients would require immediate referral to community psychiatry.
* Current or past history of meeting DSM-5 criteria for:

(the following diagnoses must have been confirmed by a qualified psychiatrist or psychologist):

* Schizophrenia;
* Psychotic Disorder (unless substance-induced or due to a medical condition);○ Borderline Personality Disorder;
* Bipolar I Disorder;
* Bipolar II Disorder;
* Other psychiatric conditions judged to be incompatible with establishment of rapport or safe exposure to psilocybin.

  * Borderline Personality Disorder, Bipolar I Disorder and Bipolar II Disorder may be considered after a psychiatric consult.
  * Bipolar I would require more in-depth investigation in relation to the history of manic episodes.

    * Meet DSM-5 criteria for Dissociative Disorder
    * Concurrent use of illicit drugs causing ongoing intoxication
    * Unstable housing conditions (homelessness)
    * First degree relatives meet DSM-5 criteria for Bipolar Disorder or Schizophrenia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1: Treatment Intervention Phase - Safety Monitoring: Adverse events (AEs), serious adverse events (SAEs) and treatment emergent adverse events (TEAEs) | Treatment intervention period: Weeks 1 through 10
  Safety in the trial will be evaluated by monitoring AEs, SAEs, and TEAEs over the 10-week intervention period. Adverse events will be defined and documented according to the adverse reporting procedures and be collected via self-report, report from others, or chart abstraction.
Primary Outcome 2: Follow-up to Treatment Phase - Safety Monitoring: Adverse events (AEs), serious adverse events (SAEs) and treatment emergent adverse events (TEAEs) | Follow-up period: Weeks 10 through 14
  Safety in the trial will be evaluated by monitoring AEs, SAEs, and TEAEs during the 30-day treatment intervention follow-up phase. Adverse events will be defined and documented according to the adverse reporting procedures and be collected via self-report, report from others, or chart abstraction.
Primary Outcome 3: Safety Monitoring: Biomedical measures - Pregnancy testing | Immediately prior to treatment intervention session (Week 5)
  A urine pregnancy test measuring beta-human chorionic gonadotropin (B-hCG) will be conducted on the pre-treatment targeted physical exam visit to ensure the participant is not pregnant. If the pregnancy test is positive, the participant will be unable to participate in the treatment intervention at Week 5 but will be invited to remain in group therapy interventions sessions (Weeks 1-10).
Primary Outcome 3: Safety Monitoring: Biomedical measures - Heart Rate | Treatment intervention session (Week 5)
  Vitals signs, including heart rate (beats per minute/BPM) will be measured before, during, and after the treatment intervention session.
Primary Outcome 3: Safety Monitoring: Biomedical measures - Blood Pressure | Treatment intervention session (Week 5)
  Vitals signs, including blood pressure (millimeters of mercury/mmHg) will be measured before, during, and after the treatment intervention session.

SECONDARY OUTCOMES:
Feasibility Outcome 1: Attendance during study intervention. | Weeks 1-10
  Feasibility outcomes will be measured using standardized assessments of treatment retention (i.e., partucipant attendance) Treatment retention will be defined as attendance in 80 % of the CoP group therapy sessions (>2 consecutive sessions) and attendance at the Week 5 psilocybin therapy session.
Feasibility Outcome 2: Post-treatment intervention Qualitative Survey | End of treatment intervention period: Week 10
  Upon completing the 10-week intervention period, all participants will complete the Roots to Thrive (RTT)-Psychedelic Assisted Therapy (PAT) Global QI Survey by answering seven (7) standard questions. Each participant will answer the same 7 questions. This survey will be administered by a member of the study team, and each question will be completed by the participant via online entry.

OTHER OUTCOMES:
Exploratory Outcome 1: Efficacy outcomes via self-report questionnaires: Adverse Childhood Events Questionnaire (ACE) | -28 to day 1 of programming (Week 0-1) and once again during Follow-up period (Weeks 10 through 14)
  The Adverse Childhood Experience (ACE) Questionnaire is a widely used validated scale with 10-item self-report measures to identify how adverse childhood experiences such as abuse and neglect may impact one's life and development. The questionnaire assesses five personal types of childhood trauma and five are related to family members. The ACE will be administered at the Baseline study visit.
Exploratory Outcome 2: Efficacy outcomes via self-report questionnaires: Patient Health Questionnaire - 9 (PHQ-9) | -28 to day 1 of programming (Week 0-1) and once again during Follow-up period (Weeks 10 through 14)
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used validated scale that is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders to measure severity of
  depression and response to treatment. The PHQ-9 will be administered at Baseline, Week 10 -Week 14 timepoints.
Exploratory Outcome 3: Efficacy outcomes via self-report questionnaires: Generalized Anxiety Disorder - 7 (GAD-7) | -28 to day 1 of programming (Week 0-1) and once again during Follow-up period (Weeks 10 through 14)
  The Generalized Anxiety Disorder-7 (GAD-7) is a widely recognized validated self-report measure scale consisting of items reflecting the symptom DSM criteria for generalized anxiety disorder and from existing anxiety scales to understand one's experience of generalized anxiety at Baseline, Week 10 -Week 14 timepoints.
Exploratory Outcome 4: Efficacy outcomes via self-report questionnaires: McGill Quality of Life Questionnaire - Extended (MQOL-E) | -28 to day 1 of programming (Week 0-1) and once again during Follow-up period (Weeks 10 through 14)
  The Generalized Anxiety Disorder-7 (GAD-7) is a widely recognized validated self-report measure scale consisting of items reflecting the symptom DSM criteria for generalized anxiety disorder and from existing anxiety scales to understand one's experience of generalized anxiety at Baseline, Week 10 -Week 14 timepoints.
Exploratory Outcome 5: Efficacy outcomes via self-report questionnaires: Watts Connectedness Scale (WCS) | -28 to day 1 of programming (Week 0-1) and once again during Follow-up period (Weeks 10 through 14)
  The Watts Connectedness scale is a new three-dimensional index of felt connectedness that measures the various aspects of connectedness such as connection to 'self', 'others', and 'world'. This validated self-report measure seeks to understand one's experience of connection. The WCS will be administered at Baseline, Week 10 -Week 14 timepoints.
Exploratory Outcome 6: Efficacy outcomes via self-report questionnaires: Substance Use & Coping Behaviours Questionnaire | -28 to day 1 of programming (Week 0-1) and once again during Follow-up period (Weeks 10 through 14)
  Participants will complete a brief series of questions around substance use and coping patterns including yes/no response options, type, frequency of various coping and substance use behaviours. This brief questionnaire will be administered at Baseline, Week 10-Week 14 study visit timepoints.